CLINICAL TRIAL: NCT04493346
Title: Shear Wave Elastography of the Liver and Predictions of Morbidity and Mortality in Subjects Undergoing Advanced Heart Failure Therapy
Brief Title: Shear Wave Elastography
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 018-164
Record Dates: First submitted 2020-07-13; First posted 2020-07-30 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure; Transplant; Failure, Heart; Decompensated Heart Failure; Fibrosis, Liver; Cirrhosis, Liver
MeSH Terms: conditions — Heart Failure; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In individuals needing a left ventricular assist device (LVAD), right heart failure (RHF) is a serious complication post-surgery, associated with worsened outcomes including mortality. However, predictors of decompensation after LVAD are not well established. Liver dysfunction pre-LVAD has been shown to be associated with poor outcomes post-LVAD, but the interplay between liver abnormalities and RHF post-LVAD is not well characterized. Liver stiffness (LS) is a measure associated with certain types of liver abnormalities (e.g., liver fibrosis; cirrhosis).

Thus, we hypothesize that elevated LS measured by SWE is associated with increased morbidity and mortality in patients undergoing LVAD implantation and yields increased need for advanced postoperative HF therapies including the use of right ventricular assist devices (RVAD) for the management of RHF.

DETAILED DESCRIPTION:
PRESTUDY ASSESSMENTS Note: Assessments that are part of the standard of care and obtained within 3-4 weeks of prestudy assessment visit, are acceptable as part of the screening tests. Results of such tests will be acceptable even if obtained prior to the execution of the Informed Consent.

Prior to entry into the study, the following assessments will be performed to determine if patient is eligible to continue in the study as per section 4.2 and 4.3 describing the inclusion and exclusion criteria for the study.

1. A signed Patient Informed Consent Form must be obtained.
2. A signed Patient Authorization Form (HIPAA) must be obtained.
3. It has been confirmed that the patient meets all inclusion criteria and none of the exclusion criteria.
4. Assessment of concomitant medications must be obtained within 4 weeks prior to registration.

ASSESSMENTS DURING STUDY

The following evaluations will be performed during the study:

1. An assessment of liver stiffness will be performed by shear wave elastography using a Supersonic Imagine Aixplorer ShearWave™ ultrasound machine. Liver stiffness assessment will be performed at a baseline visit (i.e., before LVAD placement for those undergoing LVAD therapy), and if feasible at 1 month and 6 months post-therapy (for those undergoing advanced therapy [i.e., LVAD or transplant]) or at 1 month and 6 months post-baseline (for those not undergoing advanced therapy.) FOLLOW UP ASSESSMENTS The duration of patient participation in the study will be a total of 12 months, which is counted from LVAD placement (or from baseline, for those not undergoing LVAD therapy). Follow-ups will be performed at 1 month, 6 months, and 12 months, during which the following information will be documented on the CRF.

Note: Patients who die or withdraw consent are considered off study and no further information will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients ≥18 years of age.
* Patient must be diagnosed with HF.
* Patient must be referred for an evaluation for advanced HF therapy (i.e., LVAD or heart transplantation).
* Patient must be accessible for treatment and follow-up.
* Outpatients only
* All patients must be able to understand the investigational nature of the study and give written informed consent prior to study entry.

Exclusion Criteria:

* Severe obesity (body mass index [BMI] >35 kg/m2) or severe abdominal obesity
* History of chronic or acute liver disease.
* Positive test for hepatitis C antibody or hepatitis B surface antigen reactivity
* History of intravenous drug or heavy alcohol use
* Patients with ultrasound data showing liver surface nodularity as a surrogate for advanced fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study participants are all adult patients in consideration for advanced HF therapy.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Liver stiffness (LS) measurements with development of post-LVAD RHF. | 24 months
  An assessment of liver stiffness will be performed by shear wave elastography using a Supersonic Imagine Aixplorer ShearWave™ ultrasound machine.

SECONDARY OUTCOMES:
30 day in-hospital mortality rate | 30 days
  We will perform logistic regression to determine the optimal cutpoint of LS to predict mortality at a given time point, provided the sample size is adequate.
1 year mortality rate | 1 year
  We will perform logistic regression to determine the optimal cutpoint of LS to predict mortality at a given time point, provided the sample size is adequate.

CONTACTS AND LOCATIONS:
Overall Officials: Amarinder Bindra, MD, Principal Investigator — BSWHRI
Locations (1):
- Baylor Scott & White Health research institute, Dallas, Texas, United States